CLINICAL TRIAL: NCT06167915
Title: A Randomized, Blinded, Placebo-Controlled, Dose Escalation Phase 1 Trial of Recombinant COVID-19 Trivalent (XBB.1+BQ.1.1+Prototype) Protein Vaccine （CHO Cell）（LYB002V14） in Booster Vaccination in Participants Aged 18 Years Old and Above
Brief Title: Safety and Immunogenicity of Recombinant COVID-19 Trivalent Protein Vaccine （CHO Cell）LYB002V14 in Booster Vaccination
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangzhou Patronus Biotech Co., Ltd. (Industry)
Collaborators: Yantai Patronus Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: LYB002V14/CT-CHN-101
Record Dates: First submitted 2023-12-11; First posted 2023-12-13 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: SARS-CoV-2; COVID-19 Vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low dose vaccine group (Experimental): 30μg dose of LYB002V14 vaccine IM, on day 0.
  Interventions: Biological: 30μg dose of LYB002V14
- High dose vaccine group (Experimental): 60μg dose of LYB002V14 vaccine IM, on day 0.
  Interventions: Biological: 60μg dose of LYB002V14
- Placebo group (Placebo Comparator): placebo IM, on day 0.
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: 30μg dose of LYB002V14 — 30μg dose of LYB002V14 vaccine IM, on day 0
  Arms: Low dose vaccine group
Biological: 60μg dose of LYB002V14 — 60μg dose of LYB002V14 vaccine IM, on day 0
  Arms: High dose vaccine group
Biological: placebo — placebo IM, on day 0
  Arms: Placebo group

SUMMARY:
This is a randomized, blinded, and dose escalation phase I trial in males and non-pregnant females, starting at 18 years of age, inclusive, who are in good health and meet all eligibility criteria. This clinical trial is designed to assess the safety and immunogenicity of Recombinant COVID-19 Trivalent (XBB.1+BQ.1.1+Prototype) Protein Vaccine （CHO Cell）（LYB002V14）.

DETAILED DESCRIPTION:
The study is a randomized, blinded and dose escalation Phase I clinical trial. It will evaluate the safety and immunogenicity of 2 dose levels of recombinant COVID-19 trivalent (XBB.1+BQ.1.1+Prototype) protein vaccine （CHO Cell）（LYB002V14）in booster vaccination. Approximately 120 participants aged 18 years and older will be enrolled in this study. The subjects in each dose group will randomly receive an intramuscular （IM） injection of experimental vaccine or placebo on Days 0 in the deltoid muscle at 2:1 and will be followed through 12 months post vaccination.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 18 years and above when screening.
2. Participate voluntarily and sign an informed consent form and have the ability to understand research procedures.
3. Negative SARS-CoV-2 nucleic acid test and SARS-CoV-2 IgM test.
4. Axillary body temperature is less than 37.3 degree centigrade on the day of enrollment.
5. Without a history of SARS-CoV-2 infection or known SARS-CoV-2 infection more than 3 months prior to screening.
6. Fertile women take effective contraceptive measures 1 month before enrollment; Fertile women (except those received hysterectomy, bilateral oophorectomy, tubal ligation/salpingectomy) and men of childbearing potential voluntarily agree to take effective contraceptive measures from screening to 3 months after vaccination and without a plan of pregnancy and germ cell donation.

Exclusion Criteria:

1. Have a known allergy, hypersensitivity, or intolerance to the planned investigational vaccine including any excipients of the vaccine. Have a known anaphylactic shock and other serious adverse events to other vaccine.
2. Have a known history of SARS and MERS.
3. Administration of antipyretics, painkillers or anti-allergy drugs within 24 hours prior to enrolment.
4. Receipt of subunit and/or inactivated vaccine within 7 days prior to vaccination or receipt of any live attenuated vaccine within 14 days prior to vaccination.
5. History of SARS-CoV-2 vaccination within 3 months prior to enrollment; Participants who received any immunoglobulin or blood products in the previous 3 months before enrollment, or plan to receive similar products during the study.
6. Participants with the following diseases: ①Any acute diseases or acute attacks of chronic diseases within 7 days prior to enrolment. ②Congenital malformations or developmental disorders, genetic defects, severe malnutrition, etc. ③Congenital or acquired immunodeficiency or autoimmune disease, or long-term receipt (>14 immunosuppressive agents within the past 6 months with exception of inhaled or topical steroids, or short-term use （≤14 consecutive days） of oral corticosteroids. ④Currently suffering from or diagnosed with infectious diseases, or positive screening results for human immunodeficiency virus antibody. ⑤History or family history of neurological disorders (convulsions, epilepsy, encephalopathy, etc.) or psychiatric disorders. ⑥Asplenia, or functional asplenia. ⑦Presence of severe, uncontrollable or hospitalized cardiovascular diseases, diabetes, blood and lymphatic diseases, immune diseases, liver and kidney diseases, respiratory diseases, metabolic and skeletal diseases, or malignant tumors. ⑧Contraindications to IM injections and blood draws, such as coagulation disorders, thrombotic or bleeding disorders, or conditions that needs continuous anticoagulant usage. ⑨Hypertension not controlled by medication (on-site measurement: systolic blood pressure ≥ 160mmHg and / or diastolic blood pressure ≥ 100mmHg).
7. Have a history of major surgery within 3 months before enrollment （based on the judgment of the researchers）, or has not yet fully recovered from the surgery, or has a major surgical plan during the study.
8. Those participating or planning to participate in other clinical trials during the study period.
9. Those unsuitable for participating in the clinical trial as determined by the investigator because of other abnormalities that are likely to confuse or confound the study results, or non-conformance with the maximal benefits of the participants.
10. Exclusion criteria for selected populations: those who are pregnant or breast-feeding or women of childbearing potential have a positive pregnancy test prior to vaccination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-12-26 (Estimated); Primary Completion 2024-12-26 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events and adverse reactions | Day 0 to Day 7
  Statistical description of solicited and unsolicited adverse events （AEs） will be listed. Frequencies and percentages of AEs, including overall AEs, AEs related to vaccination, AEs classified as grade 3 or worse, AEs classified as grade 3 or worse that related to vaccination, AEs leading to participant's withdrawal, AEs leading to participant's withdrawal that related to vaccination will be presented. Fisher's exact test will be used to compare the differences between the groups.

SECONDARY OUTCOMES:
Adverse events and adverse reactions | Day 0 to Day 28
  Statistical description of solicited and unsolicited adverse events （AEs） will be listed. Frequencies and percentages of AEs, including overall AEs, AEs related to vaccination, AEs classified as grade 3 or worse, AEs classified as grade 3 or worse that related to vaccination, AEs leading to participant's withdrawal, AEs leading to participant's withdrawal that related to vaccination will be presented. Fisher's exact test will be used to compare the differences between the groups.
Serious Adverse Events （SAEs） and Adverse Events of Special Interest （AESI） | Day 0 to Month 12
  Statistical description of Serious Adverse Events （SAEs） and Adverse Events of Special Interest （AESI） will be listed. Frequencies and percentages of SAEs and AESI, related to vaccination will be followed during the whole observation.
Laboratory test and vital signs related adverse events. | Day 0 to Day 3
  Indicator of Laboratory test and vital signs related adverse events will be evaluated with three days after booster vaccination.
Geometric mean titer （GMT）, Geometric Mean Fold Rise （GMFR） and seroconversion rate （SCR） of neutralizing antibodies （nAb） against variants of concern circulating during the trial. | Day 14、Day 28、Month 3 and Month 6
  The Seroconversion （SCRs） with Clopper-Pearson 95% CIs of neutralizing antibodies （Nabs） against circulating VOCs using Vesicular stomatitis virus （VSV）-based pseudovirus neutralizing assays, at Day 14、Day 28、Month 3 and Month 6 after booster immunization will be calculated for each group, compared with the baseline.
GMT, GMFR and SCR of nAb against Omicron subvariant （XBB） | Day 14、Day 28、Month 3 and Month 6
  The Seroconversion （SCRs） with Clopper-Pearson 95% CIs of neutralizing antibodies （Nabs） against Omicron subvariant （XBB） using Vesicular stomatitis virus （VSV）-based pseudovirus neutralizing assays, at Day 14、Day 28、Month 3 and Month 6 after booster immunization will be calculated for each group, compared with the baseline.
Geometric Mean Concentration （GMC）, GMFR and SCR of SARS-CoV-2 Spike protein binding antibody. | Day 14、Day 28、Month 3 and Month 6
  Geometric Mean Concentration（GMC）, GMFR and SCR with Clopper-Pearson 95% CIs of S protein-binding antibodies using ELISA assays, at baseline, at Day 14、Day 28、Month 3 and Month 6 after the booster immunization will be calculated for each group, compared with the baseline.
Th1 and Th2 cytokine responses | Day 14 and Month 6
  The counts of spot forming cells （SFCs） per 3×10^5 peripheral blood mononuclear cells （PBMCs） of Cellular immunity RBD-specific IFN-γ and IL-4 cytokine levels at baseline, Day 14 and Month 6 after booster vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Qin Yu, Master, Principal Investigator — West China Second University Hospital
Locations (1):
- West China Second University Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No